CLINICAL TRIAL: NCT00194259
Title: Sleep Apnea in Look AHEAD (Action for Health in Diabetes)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Temple University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: HL70301; NCT00350740 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2008-01

CONDITIONS: Obstructive Sleep Apnea; Type 2 Diabetes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva Samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will assess the effects of weight loss on sleep-disordered breathing (SDB) in 120 obese, type 2 diabetics with obstructive sleep apnea (OSA) from four Look AHEAD sites. Changes in SDB will be compared between subjects randomized to weight loss (Lifestyle Intervention Group) versus non-weight loss (Diabetes Education and Support Group) conditions within the context of the Look AHEAD Study. Weight loss is frequently recommended for obese patients with OSA, but the empirical foundation for this recommendation is not well substantiated. Weight loss in obese apneics improves but does not eliminate SDB. Moreover, the degree of improvement is not correlated with the amount of weight loss. This study will assess SDB before treatment and at 1 and 2 years. We will also investigate clinical measures of fat distribution that may mediate the non-linear relationship between weight loss and improvements in SDB. Finally, we will examine the role of SDB in mediating changes in blood pressure associated with weight loss.

DETAILED DESCRIPTION:
The duration of the study is 5 years; participants will be enrolled in the study for a total of 2 years. Recruitment will be based on the protocol set forth in the larger Look AHEAD trial that will occur in 8 treatment waves, spaced approximately 4 months apart. Each of these waves at the Penn site will include 40 people, making the potential subject pool approximately 320 persons.

Participants at the Penn site will be approximately 44 men and women, between 45 and 75 years of age, with a body mass index (BMI) > 25 kg/m2. All subjects will be obese type 2 diabetics who have been randomly assigned to the Lifestyle Intervention Group or the Diabetes Education and Support Group in the Look AHEAD Study. Therefore, the inclusion and exclusion criteria are determined by the parent study. Patients who are currently being treated for OSA (e.g., continuous positive airway pressure) or who have had surgical treatment for OSA will be excluded. Patients who have been previously diagnosed with OSA but are not being treated will be included. These 44 individuals represent a subset of the approximately 320 persons who will be treated at the University of Pennsylvania site.

As part of the baseline visit (before randomization) for the Look AHEAD study, Look AHEAD participants will be asked to sign a consent form for screening. Consenting participants will complete the Multivariate Apnea Prediction Form. The MAP includes weight, height, age and 3 questions about sleep-related symptoms. After the prescreen consent has been completed, the Research Coordinator will invite the participant to complete the consent form for this study. Interested subjects will be scheduled to meet with this study's Research Coordinator during the subject's next scheduled Look AHEAD visit. Participants wishing to enroll will undergo the baseline assessments and be scheduled for their baseline sleep study. Subjects will be paid $50 for this sleep assessment. After completion of the baseline sleep study, the results will be analyzed. Thirty subjects with a baseline RDI > 15 and 28 subjects with an RDI between 5 and 15 (5 < RDI < 15) will continue in the study, undergoing the same assessments at years 1 and 2.

Obstructive sleep apnea (OSA) is a syndrome characterized by frequent cessations of airflow during sleep (despite continued respiratory effort) that are caused by the closure of the pharyngeal airway. The most frequently used metric to describe OSA is the respiratory disturbance index (RDI) (sometimes referred to as the apnea-hypopnea index or AHI). RDI is defined as the average number of apnea/hypopnea events per hour of sleep. The medical consequences of OSA include an increased risk of hypertension, stroke, myocardial infarction, and premature mortality. The behavioral and psychosocial consequences of OSA include excessive daytime sleepiness, depression, sexual dysfunction, and a 3-7 fold increase in the risk of motor vehicle accidents. Among 30 to 60 year olds, 9% of women and 24% of men in the general population have an RDI > 5. The serious consequences and high prevalence of OSA clearly constitute a major public health problem.

OSA is strongly related to obesity, an important public health problem in its own right. In a series of 1000 OSA patients, two thirds had body weights > 30% above recommended. Several studies have identified body mass index (BMI) as the strongest predictor of RDI. Data from the Wisconsin Sleep Cohort Study revealed that a one standard deviation increase in BMI was associated with a four-fold increase in the risk of having an RDI > 5. Among obese patients seeking weight loss treatment, nearly 40% exhibited evidence of SDB, and 10% required treatment for OSA. The link between obesity and SDB is further supported by data showing that weight loss significantly improves SDB in obese patients with OSA. Perhaps the most compelling data about the effects of weight change on SDB, particularly weight gain, come from a very recent study of the Wisconsin Sleep Cohort that examined changes in weight and SDB over 4 years in a community sample of 690. On average, the sample experienced a 3 kg weight gain and 1.4/hr increase in RDI. Across the entire sample, on average, a 1% change in body weight was associated with a 3% change in RDI. Participants who reduced body weight by 10% experienced a 26% reduction in RDI, while those who increased body weight by 10% experienced a 32% increase in RDI. A 10% weight gain was associated with a 6-fold increase in the risk of developing a RDI > 15. These descriptive, longitudinal data are suggestive of the benefits of weight loss on SDB, but several factors limit conclusions about the effects of weight loss on obese OSA patients. First, the initial mean RDI was 4.1, so very few subjects (n = 46) had moderate or severe OSA (RDI > 15). Further, only a small number of subjects (n = 61) lost > 5% of initial body weight. Finally, similar to the broader literature on the effects of weight loss, this study is limited by the lack of a no-weight loss control group and the inability to distinguish intentional from non-intentional weight loss.

Weight loss is a frequently recommended treatment for obese patients with OSA, but the data to support this recommendation are not available. The lack of randomized trials, the study of predominantly male samples, and the absence of follow-up evaluations leave physicians and patients unsure about the clinical utility of weight loss for obese OSA patients. This study will assess the effects of weight loss on sleep-disordered breathing (SDB) in obese, type 2 diabetics with OSA (RDI > 15) who will be randomly assigned to the Lifestyle Intervention Group or the Diabetes Education and Support Group conditions as part of the larger Look AHEAD trial. Our assessment of patients at baseline, and 1 and 2 years will allow us to examine the relationship between weight change and SDB over time. We will also examine the role of neck and abdominal fat distribution in mediating the effects of weight loss on SDB. Finally, we will assess the impact of SDB in mediating changes in blood pressure associated with weight loss.

All subjects will be obese type 2 diabetics who are enrolled in the larger Look AHEAD Study. Fifty-eight subjects in total will be needed. Thirty of these subjects will have an RDI > 15 and 28 subjects will have an RDI of 5-14.9 and all will have been randomized to either the Lifestyle Intervention Group or the Diabetes Education and Support Group.

All participants will complete the following assessments:

Nocturnal polysomnography (PSG). Overnight, unattended PSGs will be recorded in participants' homes using the Compumedics' PS2 portable sleep system. Two sleep technicians will go to the participant's home at 8:00-9:00 PM on the night of the PSG. A series of calibrations will be performed and signal quality and sensor positions will be adjusted as necessary. Before the technicians depart, the device will be set to activate 60 minutes prior to the subject's intended bedtime. The subject will then be asked to sit quietly and read or watch television for the duration of the time until lights out at his/her regular bedtime. The next morning, the 2 sleep technicians will return to the participant's home to remove the electrodes and sensors and to retrieve the equipment.

Neck circumference. Neck fat distribution will be estimated by a measurement of the neck circumference at baseline and at 1 and 2 years by this study's Research Coordinator at the Look AHEAD annual clinic visit. All measurements will be performed twice and recorded to the nearest 0.1 cm.

Blood pressure. Blood pressure will be assessed at baseline and at years 1 and 2 in the participant's home by the sleep technician. Measurements will be taken at night before the equipment is attached and in the morning after the equipment has been detached. Since the PSG is anchored to the participants usual sleep and wake schedule, we will obtain a morning and evening blood pressure at approximately the same times of day. Blood pressure will be measured in the dominant arm after 5 minutes of quiet rest in a seated position. Two measurements, separated by 1 minute, will be performed and averaged.

Sagittal diameter. Sagittal diameter will be measured by the Holtain-Kahn Abdominal Caliper at baseline and at 1 and 2 years by the Research Coordinator at the Look AHEAD annual clinic visit. The measurement will be performed twice and recorded to the nearest 0.1 cm.

Questionnaires. Daytime sleepiness will be assessed by the Epworth Sleepiness Scale (ESS). The ESS is a self-administered questionnaire measuring the general level of daytime sleepiness. The ESS significantly distinguishes patients with and without OSA; a score above 10 is considered indicative of pathological sleepiness. Furthermore, it has been shown to decrease for OSA patients treated with continuous positive airway pressure (CPAP). Quality of life specific to sleep apnea will be assessed by the Functional Outcomes of Sleep Questionnaire (FOSQ). The FOSQ is a measure assessing the impact of disorders of excessive sleepiness on functional outcomes relevant to daily behaviors and quality of life. The FOSQ reliably distinguishes apneics and controls and is sensitive to treatment effects. These measures will be assessed at baseline and at 1 and 2 years by this study's Research Coordinator at the Look AHEAD clinic visits and should take approximately 10 minutes to complete.

Upper airway assessment. A brief (< 10 minutes) standardized clinical assessment of upper airway and craniofacial features that distinguishes apneics and non-apneics will be performed at baseline and at years 1 and 2 by the Research Coordinator.

Sleep log. Participants will be given a sleep log to keep for 7 days prior to their in-home sleep study. Each morning when they wake up and each evening before going to bed they will answer a few questions concerning the quality of their sleep and their daytime activities.

The procedures and treatments proposed in this study pose few known risks to subjects' physical and psychological well-being. The requirements imposed upon participants for this ancillary study pose no additional risks than those already present in the larger Look AHEAD trial. There are no invasive measures associated with this study.

The benefits to the subjects studied in this research protocol, and to society at large, far surpass the risks. Our study will provide valuable sleep assessments to a population at high risk for sleep apnea, a significant benefit since most cases of SDB in the United States (90%) are undetected. Furthermore, our study will offer both patients and their physicians valuable information necessary in making subsequent decisions regarding the clinical management of any SDB. The requirements imposed upon participants for this ancillary study pose no additional risks than those already present in the larger Look AHEAD trial.

Although weight loss is a frequently recommended treatment for obese patients with OSA, there has only been one randomized controlled trial including a no weight loss group. Therefore, findings from this study will provide important information to society at large in determining the effectiveness of weight loss treatment for OSA, a serious health problem.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in LookAhead
* Type II Diabetes and Sleep Apnea

Exclusion Criteria:

* Determined by parent study, LookAhead

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type II diabetes previously enrolled into the "Look-AHEAD" Study. Comid diagnosis of sleep apnea
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2001-08; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Effects of OSA on weight | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Foster, Ph.D., Principal Investigator — Temple University; Richard Millman, M.D., Principal Investigator — Brown University; Mark Sanders, AB, MD, FCCP, D'ABSM, Principal Investigator — University of Pittsburgh; Gary Zammit, Ph.D., Principal Investigator — St. Luke's-Roosevelt Hospital Center; Samuel T Kuna, M.D., Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - St. Luke's Roosevelt Hospital, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island

REFERENCES:
- [Derived] Shechter A, Foster GD, Lang W, Reboussin DM, St-Onge MP, Zammit G, Newman AB, Millman RP, Wadden TA, Jakicic JM, Strotmeyer ES, Wing RR, Pi-Sunyer FX, Kuna ST; Sleep Ahead Research Group of the Look Ahead Research Group. Effects of a lifestyle intervention on REM sleep-related OSA severity in obese individuals with type 2 diabetes. J Sleep Res. 2017 Dec;26(6):747-755. doi: 10.1111/jsr.12559. Epub 2017 May 31. PMID 28560832
- [Derived] Kline CE, Reboussin DM, Foster GD, Rice TB, Strotmeyer ES, Jakicic JM, Millman RP, Pi-Sunyer FX, Newman AB, Wadden TA, Zammit G, Kuna ST; Sleep AHEAD Research Group of the Look AHEAD Research Group. The Effect of Changes in Cardiorespiratory Fitness and Weight on Obstructive Sleep Apnea Severity in Overweight Adults with Type 2 Diabetes. Sleep. 2016 Feb 1;39(2):317-25. doi: 10.5665/sleep.5436. PMID 26446118
- [Derived] Shechter A, St-Onge MP, Kuna ST, Zammit G, RoyChoudhury A, Newman AB, Millman RP, Reboussin DM, Wadden TA, Jakicic JM, Pi-Sunyer FX, Wing RR, Foster GD; Sleep AHEAD Research Group of the Look AHEAD Research Group. Sleep architecture following a weight loss intervention in overweight and obese patients with obstructive sleep apnea and type 2 diabetes: relationship to apnea-hypopnea index. J Clin Sleep Med. 2014 Nov 15;10(11):1205-11. doi: 10.5664/jcsm.4202. PMID 25325608
- [Derived] Foster GD, Borradaile KE, Sanders MH, Millman R, Zammit G, Newman AB, Wadden TA, Kelley D, Wing RR, Pi-Sunyer FX, Reboussin D, Kuna ST; Sleep AHEAD Research Group of Look AHEAD Research Group. A randomized study on the effect of weight loss on obstructive sleep apnea among obese patients with type 2 diabetes: the Sleep AHEAD study. Arch Intern Med. 2009 Sep 28;169(17):1619-26. doi: 10.1001/archinternmed.2009.266. PMID 19786682
- [Derived] Foster GD, Sanders MH, Millman R, Zammit G, Borradaile KE, Newman AB, Wadden TA, Kelley D, Wing RR, Sunyer FX, Darcey V, Kuna ST; Sleep AHEAD Research Group. Obstructive sleep apnea among obese patients with type 2 diabetes. Diabetes Care. 2009 Jun;32(6):1017-9. doi: 10.2337/dc08-1776. Epub 2009 Mar 11. PMID 19279303